CLINICAL TRIAL: NCT03996889
Title: Treatment of Popliteal Aneurysms With VIABAHN Stent Graft in Elective Surgery: Multicenter Prospective Registry of the Research in Vascular Surgery University Association (AURC)
Brief Title: Treatment of Popliteal Aneurysms With VIABAHN Stent Graft in Elective Surgery
Acronym: VAP-AURC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: VAP-AURC
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Popliteal Aneurysm
MeSH Terms: conditions — Popliteal Artery Aneurysm | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Popliteal aneurysm patients with GORE VIABAHN®: The study population will include all popliteal aneurysm patients treated with GORE VIABAHN® stent graft in scheduled elective surgery, whether symptomatic or asymptomatic.
  Interventions: Device: Endovascular treatment of aneurysms of the popliteal artery by GORE VIABAHN® stent in elective surgery

INTERVENTIONS:
Device: Endovascular treatment of aneurysms of the popliteal artery by GORE VIABAHN® stent in elective surgery — The intervention can be performed under local anesthesia (LA), regional locus (ALR) or general anesthesia (AG) (data collected) by first approach: percutaneous or conventional.
  The data collected are:
  * Number of GORE VIABAHN® stent used (length and diameter of each)
  * Embolization of collaterals and other related actions
  * Operative complications
  * Intraoperative fibrinolysis
  * Collar cover> 2 cm
  * Lack of overlap in the "overlap zone" (nb: between 4 and 8 cm above the joint spacing)
  * Arteriography in profile, kink

SUMMARY:
This multicentric, prospective study will evaluate the medium-term outcomes of patients implanted with GORE VIABAHN® stent grafts for popliteal artery aneurysms in scheduled elective surgery with the registry of the Research in Vascular Surgery University Association (AURC)

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old at time of treatment
* symptomatic or asymptomatic popliteal artery aneurysm needing surgery
* scheduled elective surgery

Exclusion Criteria:

* life expectancy of <1 year
* thrombotic occlusion of popliteal artery
* intolerance to antiplatelet drugs (antiaggregants)
* known allergies to GORE VIABAHN® stent graft materials/composition
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all popliteal aneurysm patients treated with GORE VIABAHN® stent graft in scheduled elective surgery, whether symptomatic or asymptomatic.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Major limb events | 2 years of follow-up
  Composite criterion associating Target Lesion Revascularization (TLR) and Rate of major amputation.
  An Echo-Doppler imaging examination will be performed and the following parameters and information should be collected:
  * Permeability
  * Intra-stent restenosis
  * Systolic pressure index

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital pneumologique et cardiovasculaire Louis Pradel (HCL), Bron, France